CLINICAL TRIAL: NCT01053858
Title: Triamcinolone or Bevacizumab for Central Retinal Vein Occlusion With Poor Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009_10_12
Record Dates: First submitted 2010-01-14; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Central Retinal Vein Occlusion With 20/200 or Worse Visual Acuity
Keywords: bevacizumab,triamcinolone, intravitreal injection
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bevacizumab (Active Comparator): intravitreal bevacizumab or triamcinolone determined by single physician
  Interventions: Procedure: intravitreal injection
- triamcinolone (Active Comparator)
  Interventions: Procedure: intravitreal injection

INTERVENTIONS:
Procedure: intravitreal injection — intravitreal bevacizumab( 1.25 mg) or triamcinolone( 4mg) injection

SUMMARY:
To evaluate the effect of intravitreal bevacizumab with intravitreal triamcinolone for the treatment of central retinal vein occlusion (CRVO) presenting poor visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* central macular thickness of more than 250 μm and baseline visual acuity of 20/200 or worse than 20/200 in patient with central retinal vein occlusion

Exclusion Criteria:

* previous treatment such as intravitreal injection, subtenon injection, or laser photocoagulation since the time of onset
* Patients with a history of glaucoma, neovascular glaucoma, diabetic retinopathy, and macular disorders
* neovascularization on the disc or elsewhere or rubeosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity | baseline, 1 month, 2 months, 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
central macular thickness by optical coherence tomography | baseline, 1 month, 2 months, 3 months, 6 months 12months

CONTACTS AND LOCATIONS:
Locations (1):
- keoung ik Na, Chuncheon, anyang, South Korea